CLINICAL TRIAL: NCT04641871
Title: An Exploratory, Open-label, Multicenter Phase 1b Trial to Evaluate Safety and Efficacy of Sym021 (Anti-PD 1) in Combination With Either Sym022 (Anti-LAG-3) or Sym023 (Anti-TIM-3) or Sym023 and Irinotecan in Patients With Recurrent Advanced Selected Solid Tumor Malignancies
Brief Title: Sym021 in Combination With Either Sym022 or Sym023 or Sym023 and Irinotecan in Patients With Recurrent Advanced Selected Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Symphogen A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sym021-02
Record Dates: First submitted 2020-10-29; First posted 2020-11-24 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Metastatic Cancer; Solid Tumor
Keywords: Locally advanced/unresectable; Metastatic solid tumor; Anti-PD-1; PD-1; PD1; Anti-TIM-3; TIM-3; TIM3; Cholangiocarcinoma; CCA; Biliary Tract Carcinomas; Gallbladder; Esophageal Squamous Cell Carcinoma; ESCC; Irinotecan
MeSH Terms: conditions — Neoplasm Metastasis; Cholangiocarcinoma; Esophageal Squamous Cell Carcinoma | interventions — spartalizumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sym021+Sym022 [ARM A] for BTC patients (Experimental): Sym021 will be infused over approximately 30 minutes (+10 minutes), followed by a 30-minute post-dosing interval before infusion of Sym022 over approximately 30 minutes (+10 minutes). The duration of each infusion may be extended by 30 minutes, or longer, if indicated.
  Interventions: Drug: Sym021; Drug: Sym022
- Sym021+Sym023 [ARM B] for BTC patients (Experimental): Sym021 will be infused over approximately 30 minutes (+10 minutes), followed by a 30-minute post-dosing interval before infusion of Sym023 over approximately 30 minutes (+10 minutes). The duration of each infusion may be extended by 30 minutes, or longer, if indicated.
  Interventions: Drug: Sym021; Drug: Sym023
- Sym021+Sym023+irrinotecan for BTC patients (Experimental): Sym021 will be infused over approximately 30 minutes (+10 minutes), followed by a 30-minute post-dosing interval before infusion of Sym023 over approximately 30 minutes (+10 minutes). The duration of each infusion may be extended by 30 minutes, or longer, if indicated. After another 30-minute post-dosing interval, irinotecan will be infused over 90 minutes.
  Interventions: Drug: Sym021; Drug: Sym023; Drug: Irinotecan Hydrochloride
- Sym021+Sym023+irrinotecan for ESCC patients (Experimental): Sym021 will be infused over approximately 30 minutes (+10 minutes), followed by a 30-minute post-dosing interval before infusion of Sym023 over approximately 30 minutes (+10 minutes). The duration of each infusion may be extended by 30 minutes, or longer, if indicated. After another 30-minute post-dosing interval, irinotecan will be infused over 90 minutes.
  Interventions: Drug: Sym021; Drug: Sym023; Drug: Irinotecan Hydrochloride

INTERVENTIONS:
Drug: Sym021 — IV infusion over 30 minutes on day 1 and 15 of each cycle.
  Other Names: Anti-PD-1
Drug: Sym022 — IV infusion over 30 minutes on day 1 and 15 of each cycle.
  Other Names: Anti-LAG-3
  Arms: Sym021+Sym022 [ARM A] for BTC patients
Drug: Sym023 — IV infusion over 30 minutes on day 1 and 15 of each cycle.
  Other Names: Anti-TIM-3
  Arms: Sym021+Sym023 [ARM B] for BTC patients; Sym021+Sym023+irrinotecan for BTC patients; Sym021+Sym023+irrinotecan for ESCC patients
Drug: Irinotecan Hydrochloride — IV infusion over 90 min on day 1 and 15 of the first 2 cycles. After 2 cycles of treatment, irinotecan may be discontinued at the Investigator's discretion
  Arms: Sym021+Sym023+irrinotecan for BTC patients; Sym021+Sym023+irrinotecan for ESCC patients

SUMMARY:
The study will evaluate the preliminary efficacy of 3 combinations (Sym021+Sym022, Sym021+Sym023 and Sym021+Sym023+irinotecan) in patients with biliary tract carcinomas (BTC) and with esophageal squamous cell carcinoma (ESCC) by assessing overall response rates (ORRs) per Investigator assessment using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 The study will also evaluate the safety and tolerability profile of the 3 combinations

DETAILED DESCRIPTION:
The study will evaluate safety and efficacy in patients with:

* Biliary tract carcinomas patients who have progressed on one prior line of gemcitabine and platinum-based chemotherapy in the metastatic setting.
* Esophageal squamous cell carcinoma patients who have progressed on one prior line of platinum-based chemotherapy in the metastatic setting.

The trial is set up as 3 sub-studies.

* Sub-study 1 includes biliary tract carcinoma patients and is composed of 2 investigational combination treatment arms (Sym021+Sym022 [Arm A] and Sym021+Sym023 [Arm B]).
* Sub-study 2, includes biliary tract carcinoma patients and is composed of one investigational combination treatment arm:Sym021+Sym023+irinotecan. A safety lead- in phase is included to assess tolerability of the combination. A Study Safety Team will review clinical and laboratory safety data and will make decisions regarding the continued enrollment after the safety lead-in phase.
* Sub-Study 3, includes esophageal squamous cell carcinoma patients and is composed of one investigational combination treatment arm: Sym021+Sym023+irinotecan. Dose of irinotecan in this arm will be selected based upon the safety lead in in sub-study 2 period.

August 2021 : Based upon results from a recent per protocol Interim Analysis (IA) it is has been decided as of 3rd of August 2021 to stop further enrollment into Sub-study 1 Arm A (Sym021+Sym022). Future patients will be allocated to either Sub-study 1 Arm B (Sym021+Sym023) or Sub-study 2 (Sym021+Sym023+irinotecan).

ELIGIBILITY:
Inclusion Criteria:

For Sub-study 1 and 2:

* Patients with locally advanced or metastatic biliary tract carcinoma including adenocarcinoma of the intra- and/or extra-hepatic bile ducts and gallbladder carcinoma. Patients with ampullary cancers are excluded.
* Patients must only have received and progressed on or be intolerant of first-line gemcitabine and platinum-based chemotherapy in metastatic/advanced setting and should not have received prior anti-PD-(L)1 therapy. Patients with known fibroblast growth factor receptor 2 (FGFR2) fusion or rearrangement, or isocitrate dehydrogenase 1 (IDH1) mutation will be excluded. Prior anti-PD-(L)1 therapy may be allowed during the trial if regulatory approval for such therapy is obtained while this trial is enrolling.

For Sub-study 3:

* Patients with with locally advanced or metastatic esophageal squamous cell carcinoma
* Patients must only have received and progressed on or be intolerant of first-line platinum-based chemotherapy in metastatic/advanced setting and should have received prior anti-PD-(L)1 therapy. Patients with mixed adenosquamous histology cancers are excluded.

For all Sub-studies :

* Patients with measurable disease according to RECIST v1.1
* Patients with an ECOG PS of 0 or 1, and anticipated life expectancy of ≥3 months
* Patients must have adequate organ function as indicated by laboratory values
* Adequate contraception required as appropriate

Exclusion Criteria:

* Patients with central nervous system (CNS) malignancy, untreated or unstable metastases
* Patients with significant cardiovascular disease
* Patients with

  1. Active thrombosis, or a history of deep vein thrombosis or pulmonary embolism, within 4 weeks prior to the first study drug dose
  2. Active uncontrolled bleeding or a known bleeding diathesis
* Patients with a significant pulmonary disease or condition
* Patients with a current or recent (within 6 months) significant gastrointestinal disease or condition
* Patients with Gilbert's syndrome or patients with UGT1A1*28 homozygosity (also known as UGT1A1 7/7 genotype)
* Patients with a significant ocular disease or condition
* Patients with an active, known or suspected autoimmune disease
* Patients with any other serious/active/uncontrolled infection
* Patients with a history of organ transplantation
* Patients with human immunodeficiency virus (HIV) (HIV 1/2 antibodies) or active infection with hepatitis B virus or hepatitis C virus
* Prior therapy with irinotecan
* For Sub-study 1 and Sub-study 2: Anti-PD-(L)1, anti -LAG-3* or anti-TIM-3 containing regimen, or combination with any other systemic or localized therapy or any other immuno-oncology (IO) therapies.
* For Sub-study 3: Anti-TIM-3 containing regimen, or combination with any other systemic or localized therapy or any other IO therapies (other than anti-PD-(L)1 agents).
* Patients must not be on warfarin, if they have a history of acute immune-related thrombocytopenia; patients must not be on strong cytochrome P450 (CYP) 3A4 inducers, strong CYP3A4 inhibitors, or strong UGT1A1 inhibitors.
* Patients with a known or suspected hypersensitivity to any of the excipients of formulated study drug
* Patients with unresolved >Grade 1 toxicity associated with any prior antineoplastic therapy
* Sub-study 1 and Sub-study 2: Patients with known FGFR2 fusion or rearrangement, or IDH1 mutation.
* For Sub-study 3: Patients with a history of significant toxicities associated with previous administration of immune checkpoint inhibitors that necessitated permanent discontinuation of that therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the preliminary efficacy of the combinations Sym021+Sym022, Sym021+Sym023 and Sym021+Sym023+irinotecan in patients with BTC or ESCC by assessing overall response rates (ORRs) per Investigator assessment using RECISTv.1.1 | Until disease progression or end of study, whichever comes first, assessed up to 24 months
  Objective Response Rate (ORR) per Investigator assessment of antitumor activity (based on radiological evidence per RECIST v1.1)
To evaluate the incidence, severity, and relationship of (S)AEs collected from administration of the first dose of study drug until 30 days after the last dose of the 3 combinations (Sym021+Sym022, Sym021+Sym023 and Sym021+Sym023+irrinotecan) | Through study completion up to 30 days after last dose of the three combinations
  Calculation of AE incidence will be based on the number of patients per AE category; AEs in total and sorted by frequency, AEs by relationship, SAEs in total and by relationship, Immune mediated AEs, Fatal AEs
To evaluate the AEs leading to dose interruption, dose delays, and permanent treatment stop of the 3 combinations (Sym021+Sym022 and Sym021+Sym023 and Sym021+Sym023 +irinotecan) | Through study completion up to a maximum of 24 months
  Calculation of AE incidence will be based on the number of patients per AE category ; AEs leading to dose interruption, dose delays, and permanent treatment stop

SECONDARY OUTCOMES:
Peak plasma (irinotecan) and serum( mAbs) Concentration (Cmax) of the 3 combinations (Sym021+Sym022 and Sym021+Sym023 and Sym021+Sym023+irinotecan) | First study dose and throughout the trial, up to 2 years
  Peak serum concentration (Cmax) for each mAbs in each combination.
Area under the serum concentration versus time curve (AUC) of the 3 combinations (Sym021+Sym022 and Sym021+Sym023 and Sym021+Sym023+ irinotecan) | First dose of study drug and throughout the trial, up to 2 years
  Area under the serum concentration versus time curve (AUC) for each mAbs in each combination.
Time to reach maximum concentration (Tmax) of the 3 combinations (Sym021+Sym022 and Sym021+Sym023 and Sym021+Sym023+irinotecan) | First dose of study drug and throughout the trial, up to 2 years
  Time to reach maximum concentration (Tmax) for each mAbs in each combination.
Trough concentration (Ctrough) of the 3 combinations (Sym021+Sym022 and Sym021+Sym023 and Sym021+Sym023 + irinotecan) | First dose of study drug and throughout the trial, up to 2 years
  Trough concentration (Ctrough) for each mAbs in each combination.
Plasma concentration for irinotecan and its metabolite in the combination Sym021+Sym023+ Irinotecan | First dose of study drug and throughout the trial, up to 2 years
  Plasma concentration at the end of infusion for irinotecan and its metabolite in the combination Sym021+Sym023+ Irinotecan
To confirm the RP2D of each combination | 36 month
  Confirmation of the RP2D, based on the dose-response relationship (in case more than one dose level is implemented), overall tolerability and safety profile, and the PK and pharmacodynamic data
Evaluation of Duration of Response (DOR) | Until disease progression or end of study, whichever comes first, assessed up to 24 months
  Duration of the OR will be determined from the day initial response is observed to day of progression is observed. Number and percentages of patients with documented OR will be presented.
Evaluation of Progression-Free Survival (PFS) | From first study drug dose until disease progression or end of study, whichever comes first, assessed up to 24 months
  Will be calculated as from the first study drug dose to the day progression of disease is confirmed radiological or date of death.
Evaluation of Disease Control Rate (DCR), defined as CR, PR, or stable disease (SD) ≥6 months | Until disease progression or end of study, whichever comes first, assessed up to 6 months
  Will be calculated according to standard response criteria
Evaluation of duration of response. | Until disease progression or end of study, whichever comes first, assessed up to 24 months
  Will be calculated from the day the initial response is observed to the day progression of disease is observed
Evaluation of Objective Response Rate (ORR) per Investigator assessment (based on Immunotherapeutics Response Evaluation Criteria in Solid Tumors [iRECIST]) | Until disease progression or end of study, whichever comes first, assessed up to 24 months
  Will be based on Investigators assessment on Immunotherapeutic Response Evaluation Criteria in Solid Tumors (iRECIST)
Evaluation Overall Survival (OS) | From first dose of study drug until death or latest survival follow-up assessed up to 30 month
  Overall survival will be derived from start of treatment until death or latest survival follow-up.
Evaluation of immunogenicity of each antibody drug in the combinations | From screening up to 30 months
  Occurrence of antidrug antibody (ADA) measured in serum at selected time points during the study

CONTACTS AND LOCATIONS:
Overall Officials: Nehal Lakhani, MD, Principal Investigator — START Midwest
Locations (17):
- United States (12):
  - University of Colorado, Aurora, Colorado
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - University of Kansas Medical Center (KUMC), Westwood, Kansas
  - START Midwest, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Mount Sinai - PRIME, New York, New York
  - Montefiore Medical Center PRIME, The Bronx, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - MD Anderson, Houston, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- France (2):
  - Centre Georges-François Leclerc, Department of Medical Oncology, Dijon
  - Institut de Cancerologie de L'Ouest, Saint-Herblain
- Spain (2):
  - Vall d'Hebron Institute of Oncology, Barcelona
  - Hospital Universitario San Carlos, Madrid

IPD SHARING:
Plan to Share IPD: No